CLINICAL TRIAL: NCT01167101
Title: Is Rebamipide Effective on the Healing of Iatrogenic Gastric Ulcer After Endoscopic Mucosal Resection? : Multicenter, Randomized, and Prospective Study
Brief Title: Is Rebamipide Effective on the Healing of Iatrogenic Gastric Ulcer After Endoscopic Mucosal Resection?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangdong Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Shin, Woon Geon, Professor, Kangdong Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-62
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Stomach Ulcer
Keywords: Rebamipide; gastric ulcer; healing rate; iatrogenic gastric ulcer after endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Ulcer | interventions — rebamipide; Pantoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pantoprazole (Other): controls Pantoprazole 40mg qd for 28days
  Interventions: Drug: pantoprazole
- Pantoprazole + Rebamipde (Active Comparator): Pantoprazole 40mg qd + Rebamipide 100mg Tid for 28days
  Interventions: Drug: Rebamipide; Drug: pantoprazole

INTERVENTIONS:
Drug: Rebamipide — Rebamipide 100mg Tid for 28days
  Arms: Pantoprazole + Rebamipde
Drug: pantoprazole — pantoprazole 40mg qd for 28days

SUMMARY:
Treatment strategy of post endoscopic submucosal dissection (ESD) ulcer is not yet conclusive. Rebamipide is a mucosal protective agent widely used in East Asia and has good effect on quality of ulcer healing (QOUH). The investigators will conduct this randomized controlled study to assess the effect of a combination therapy of rebamipide and proton pump inhibitor (PPI) on post ESD ulcer healing.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent ESD for gastric adenoma or cancer

Exclusion Criteria:

* subjects with previous gastric surgery
* subjects taking aspirin, anticoagulant, or antiplatelet agent
* subjects having malignancy except gastric cancer
* pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Healing efficacy of Rebamipide in the treatment of iatrogenic gastric ulcer | at 2month after endoscopic submucosal dissection (ESD)
  Healing efficacy will be assessed by the change of ulcer size. Quality of Ulcer Healing(QOUH) wil be assessed by nodularity in the healed ulcer by two endoscopist.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangdong Sacred Heart Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin WG, Kim SJ, Choi MH, Kim KO, Jang HJ, Park CH, Baek IH, Kim KH, Baik GH, Kae SH, Kim JH, Kim HY. Can rebamipide and proton pump inhibitor combination therapy promote the healing of endoscopic submucosal dissection-induced ulcers? A randomized, prospective, multicenter study. Gastrointest Endosc. 2012 Apr;75(4):739-47. doi: 10.1016/j.gie.2011.11.004. Epub 2012 Jan 26. PMID 22281110